CLINICAL TRIAL: NCT03450954
Title: Amniotic Membrane Transplant in Symptomatic Bullous Keratopathy Patients: Confocal Microscopy & AS-OCT Long Term Results
Brief Title: Long Term Results of Amniotic Membrane Transplant in Bullous Keratopathy Patients
Status: Completed | Type: Observational
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Gillian Siu, Resident Specialist, Prince of Wales Hospital, Shatin, Hong Kong
Other Study IDs: CRE-2013.687
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Bullous Keratopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case(AMT patients): patients who have undergone amniotic membrane transplant in our unit up till 2016.
  Interventions: Procedure: Amniotic membrane transplant
- Control(Patients without AMT): bullous keratopathy patients awaiting endothelial keratoplasty

INTERVENTIONS:
Procedure: Amniotic membrane transplant — Amniotic membrane graft was transplanted onto the bullous cornea by the inlay technique
  Groups: Case(AMT patients)

SUMMARY:
A retrospective study including 22 patients who have undergone amniotic membrane transplant in our unit up till 2016. Confocal microscopy and anterior segment optical coherence tomography (ASOCT) were performed to assess the retention of amniotic membrane and to detect any corneal structural changes. Comparison was made with 5 controls who had bullous keratopathy awaiting endothelial keratoplasty.

DETAILED DESCRIPTION:
This retrospective cohort study (CREC Ref No.: CRE-2013.687) was approved by the Joint Chinese University of Hong Kong-New Territories East Cluster Clinical Research Ethics Committee. All patients who had AMT done due to symptomatic bullous keratopathy at the Prince of Wales Hospital and Alice Ho Miu Ling Nethersole Hospital (from 1998 onwards till June 2016) were invited back for confocal microscopy and anterior segment optical coherence tomography (ASOCT) at the clinic by the principal investigator (GS) from October to November 2016.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have undergone amniotic membrane transplant in our cluster up till 2016.
* Patients who have bullous keratopathy on conservative treatment such as lubricants, bandage contact lens

Exclusion Criteria:

* patients who refuse to participate in the study, have passed away or cannot return for the clinical assessment will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases who have undergone amniotic membrane transplant in our unit up till 2016 and controls who had bullous keratopathy awaiting endothelial keratoplasty
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Amniotic membrane retention | from date of operation till 2016
  Amniotic membrane retention in the cornea was assessed with confocal microscopy

SECONDARY OUTCOMES:
Pain | from date of operation till 2016
  pain score (from 0-10, scale interval 1, 0 no pain, 10 most painful)reduction after amniotic membrane tranplant

CONTACTS AND LOCATIONS:
Overall Officials: Gillian DJ Siu, MBChB, Principal Investigator — The Prince of Wales Hospital

IPD SHARING:
Plan to Share IPD: No